CLINICAL TRIAL: NCT02665910
Title: A Phase I, Randomized, Placebo-Controlled, Multiple Doses Escalation Study to Investigate Safety, Pharmacokinetics and Pharmacodynamics of SHR0302 in Patients With RA
Brief Title: Multiple Doses Escalation Study of SHR0302 in Rheumatoid Arthritis (RA) Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR0302-102
Record Dates: First submitted 2016-01-24; First posted 2016-01-28 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — ivarmacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SHR0302 (Experimental): Multiple ascending doses (2, 5, 10, 25 mg), oral tablets
  Interventions: Drug: SHR0302
- SHR0302 placebo comparator (Placebo Comparator): Multiple ascending doses (2, 5, 10, 25 mg), oral tablets (matching corresponding study medication)
  Interventions: Drug: SHR0302 placebo comparator

INTERVENTIONS:
Drug: SHR0302 — Oral tablets (1 mg, 5 mg, 10 mg)
  Arms: SHR0302
Drug: SHR0302 placebo comparator — Oral tablets (1 mg, 5 mg, 10 mg) (matching corresponding study medication)
  Arms: SHR0302 placebo comparator

SUMMARY:
Condition: Rheumatoid Arthritis Intervention: Drug: SHR0302; Drug: SHR0302 placebo comparator Phase: Phase 1 Study Type: Interventional Study Design: Treatment, Parallel Assignment, Double Blind (Subject, Caregiver, Investigator, Outcomes Assessor), Randomized

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects who are 18~70 years of age on the day of signing informed consent,
* Have a diagnosis of RA meeting the 1987 ACR/EULAR criteria of RA and ACR functional class I-III,
* Body mass index (BMI = weight/height squared (kg/m2)) within the range of 19 to 30,
* Have agreed to not use any anti- rheumatic drug except for study drugs during the study period.

Exclusion Criteria:

* Current therapy with any disease modifying anti-rheumatic drug (DMARD), with the exception of Methotrexate (MTX), Leflunomide, sulfasalazine, antimalarials, gold preparations, penicillamine, which must have discontinued for a period of at least 7 t1/2s prior to dosing,
* Previous RA treatment with DMARDs or drugs with strong immunosuppressive effect in 3 months prior to dosing (12 months for rituximab or other B cell depleting agents),
* Previous therapy with NSAIDs or oral glucocorticoids in 2 weeks before dosing,
* Any parenteral (intramuscular or intravenous injection) or intra-articular corticosteroids therapy in 4 weeks before dosing,
* Previous treatment with interferons in 4 weeks before dosing.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events and the number of volunteers with adverse events as a measure of safety and tolerability. | up to 48 hrs postdose
  Tests will be performed to assess whether the study drug has any potentially adverse effect (laboratory tests on blood and urine for functioning of organs; cardiovascular testing, i.e. of heart and blood circulation). Also, participants will carefully be monitored by medical staff for vital signs, and asked to report any side effect experienced in the course of the study

SECONDARY OUTCOMES:
The maximum plasma concentration (Cmax) of SHR0302 | At protocol-specified times up to 48 hrs postdose
  Blood samples are taken on various timepoints to assess the pharmacokinetic parameters
The area under the plasma concentration-time curve (AUC) of SHR0302 | At protocol-specified times up to 48 hrs postdose
t1/2 of SHR0302 | At protocol-specified times up to 48 hrs postdose

OTHER OUTCOMES:
Pharmacodynamics (PD) parameters of percent and actual change from baseline for a panel of JAK dependent biomarkers | At protocol-specified times up to 24 hrs postdose
  To characterize the effects of SHR0302 on mechanism of action-related biomarkers in the blood over time - pharmacodynamics (PD) - in RA.

CONTACTS AND LOCATIONS:
Overall Officials: Pei Hu, PhD, Principal Investigator — Peking Union Medical College Hospital; Xiaofeng Zeng, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided